CLINICAL TRIAL: NCT05729737
Title: Prediction and Evaluation of Chemotherapy Treatment Response Using Contrast Enhanced Ultrasound in Unresected Localized Pancreatic Cancer
Brief Title: Radiographic Response to Chemotherapy in Unresected Localized Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 82171968
Record Dates: First submitted 2022-12-25; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2022-12

CONDITIONS: Pancreatic Cancer; Ultrasonography; First-line Chemotherapy
Keywords: early chemotherapy response; contrast-enhanced ultrasound
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pancreatic ductal adenocarcinoma: Patients who planned to receive first-line chemotherapy for pathologically diagnosed PDAC were recruited.
  Intervention:Diagnostic test:Contrast-enhanced ultrasound
  Interventions: Diagnostic Test: Contrast-enhanced ultrasound(CEUS)

INTERVENTIONS:
Diagnostic Test: Contrast-enhanced ultrasound(CEUS) — CEUS is a quantitative kinetic imaging modality that can assess intravascular blood flow in pancreatic tumors, it is safe and widely used in liver and pancreatic disease.

SUMMARY:
The goal of this observational study is to explore whether contrast-enhanced ultrasound (CEUS) can early predict and evaluate the treatment response of first-line chemotherapy in locally advanced and borderline resectable pancreatic cancers.

The main questions it aims to answer are:

Question 1: What quantitative parameters of CEUS performed before first-line chemotherapy can predict the early treatment response of patients with locally pancreatic cancer?Question 2: Can CEUS reflect early neovascular changes after first-line chemotherapy in pancreatic tumors? Participants will receive CEUS examination carried out by experienced operators before the first cycle of chemotherapy and after 2 treatment cycles.

DETAILED DESCRIPTION:
Pancreatic cancer is a highly fatal disease with a low 5-year survival rate of approximately 9% in the United States. Due to vague symptoms and early involvement of vessels, surgical treatment is only feasible for 20% of patients. First-line chemotherapy, which can improve the rate of R0 resection, is increasingly being used and is preferred in the ASCO guidelines for patients with locally advanced and borderline resectable pancreatic cancers. Early prediction and evaluation of the treatment response can provide prognostic information and enable oncologists to tailor therapeutic strategies.

Contrast-enhanced ultrasound (CEUS) is of interest for its ability to gain macrovascular and microvascular information about organs and to aid our understanding of the complexity of angiogenesis in different types of tumors. CEUS is a quantitative kinetic imaging modality that can assess intravascular blood flow in pancreatic tumors even at the capillary level. Our previous studies have confirmed that the enhancement patterns of CEUS in pancreatic ductal adenocarcinoma (PDAC) have correlation with the overall survival time. Now we hypothesize that the enhancement patterns before first-line chemotherapy can predict the treatment response and the changes in the pharmacokinetics of contrast material after treatment would reflect early neovascular changes in pancreatic tumors.

The investigators plan to recruit patients who are about to receive first-line chemotherapy for pathologically diagnosed PDAC from the department of General Surgery and Medical Oncology of our hospital. The patients will receive CEUS examination before the first cycle of chemotherapy and after 2 treatment cycles. Quantitative perfusion analysis will be performed by experienced radiologists and artificial intelligence for all of the images. According to the published literature, clinical response in patients were evaluated based on the Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1) combined with the changes of serum levels of CA 19-9. Changes of CEUS quantitative perfusion parameters will be compared to clinical measurement of response to treatment taking into consideration standard response criteria including radiological imaging, serum CA 19-9 levels and repeat pathology as applicable

ELIGIBILITY:
Inclusion Criteria:

* The main inclusion criteria were histologically proven pancreatic ductal adenocarcinoma and medical fitness for first-line chemotherapy Patients were consent to receive examinations of contrast enhanced ultrasound

Exclusion Criteria:

* Patients with distal metastases or patients refusing chemotherapy Patients who were not suitable for contrast-enhanced ultrasound ,such as pregnant or lactating women Patients without complete clinical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients were diagnosed as pancreatic ductal adenocarcinoma pathologically and planned to receive first-line chemotherapy. The patients could receive regular follow up.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
RECIST 1.1 Therapeutic Responses to 4 cycles | estimated to be 4 months
  The patients underwent baseline and repeat MDCT imaging (after 4 cycle). Tumor response was determined by RECIST 1.1 and was defined as a >30% reduction in tumor size as determined by the sum of the longest diameters of each index lesion.
Serum CA 19-9 Responses to 4 cycles | estimated to be 4 months
  Serum CA19-9 levels were detected before chemotherapy and at the end of Cycle 4(each cycle is 21 days). Patients with normal CA19-9(<37 U/mL) post-chemotherapy, whether normal or elevated pre-chemotherapy are defined as "Optimal CA19-9 Response".
Evaluate if tumor uptake of contrast agent is predictive of response to chemotherapy therapy measured by comparison of Peak Intensity (PI) at CEUS imaging prior to and after 2 cycles chemotherapy | Baseline and after 2 cycles of chemotherapy (estimated to be 2 months)
  Before initiation of the chemotherapy and at the end of Cycle 2 (each cycle is 21 days) of chemotherapy, patients would receive CEUS examination. The dynamic CEUS images of each lesion were analysed with the aid of time-intensity curves (TICs) drawn by QLAB software (Philips Healthcare, Andover, MA) and artificial intelligence. PI measurements will be compared to clinical measurement of response to treatment taking into consideration standard response criteria including radiological imaging, serum CA 19-9 levels and repeat pathology as applicable.
Evaluate if the time to peak (TP) is predictive of response to chemotherapy therapy measured by comparison of TP at CEUS imaging prior to the start of first-line chemotherapy and TP at imaging performed after 2 cycles chemotherapy | Baseline and after 2 cycles of chemotherapy (estimated to be 2 months)
  Before initiation of the chemotherapy and at the end of Cycle 2 (each cycle is 21 days) of chemotherapy, patients would receive CEUS examination. The dynamic CEUS images of each lesion were analysed with the aid of time-intensity curves (TICs) drawn by QLAB software (Philips Healthcare, Andover, MA) and artificial intelligence. TP measurements will be compared to clinical measurement of response to treatment taking into consideration standard response criteria including radiological imaging, serum CA 19-9 levels and repeat pathology as applicable.

SECONDARY OUTCOMES:
Assessment of overall survival | From first day of protocol examination to the date of death due to any cause and will be censored at the date of last follow-up for patients still alive up to 2 years
  Overall survival (OS) was measured from time of diagnosis to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ke Lv, MD, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Hester CA, Perri G, Prakash LR, Maxwell JE, Ikoma N, Kim MP, Tzeng CD, Smaglo B, Wolff R, Javle M, Overman MJ, Lee JE, Katz MHG. Radiographic and Serologic Response to First-Line Chemotherapy in Unresected Localized Pancreatic Cancer. J Natl Compr Canc Netw. 2022 Aug;20(8):887-897.e3. doi: 10.6004/jnccn.2022.7018. PMID 35948035
- [Background] Lee YJ, Kim SH, Kang BJ, Kim YJ. Contrast-Enhanced Ultrasound for Early Prediction of Response of Breast Cancer to Neoadjuvant Chemotherapy. Ultraschall Med. 2019 Apr;40(2):194-204. doi: 10.1055/a-0637-1601. Epub 2018 Aug 13. PMID 30103213
- [Background] Zhou T, Tan L, Gui Y, Zhang J, Chen X, Dai M, Xiao M, Zhang Q, Chang X, Xu Q, Bai C, Cheng Y, Xu Q, Wang X, Meng H, Jia W, Lv K, Jiang Y. Correlation Between Enhancement Patterns on Transabdominal Ultrasound and Survival for Pancreatic Ductal Adenocarcinoma. Cancer Manag Res. 2021 Aug 31;13:6823-6832. doi: 10.2147/CMAR.S307079. eCollection 2021. PMID 34512022
- [Background] Zimmermann C, Distler M, Jentsch C, Blum S, Folprecht G, Zophel K, Polster H, Troost EGC, Abolmaali N, Weitz J, Baumann M, Saeger HD, Grutzmann R. Evaluation of response using FDG-PET/CT and diffusion weighted MRI after radiochemotherapy of pancreatic cancer: a non-randomized, monocentric phase II clinical trial-PaCa-DD-041 (Eudra-CT 2009-011968-11). Strahlenther Onkol. 2021 Jan;197(1):19-26. doi: 10.1007/s00066-020-01654-4. Epub 2020 Jul 7. PMID 32638040